CLINICAL TRIAL: NCT00106613
Title: An Exploratory Phase II, Multicenter, Open-label Trial Evaluating the Activity and Tolerability of FK228 in Patients With Metastatic Renal Cell Carcinoma That is Progressive Following or During Immunotherapy
Brief Title: A Research Study for Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJ-228-0001; NCT00058630 (obsolete NCT alias); NCT00060216 (obsolete NCT alias)
Record Dates: First submitted 2005-03-28; First posted 2005-03-29 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Carcinoma, Renal Cell; Neoplasm Metastasis
Keywords: Renal Cell Carcinoma; Metastatic Cancer; Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FK228 (romidepsin) (Experimental): 13 mg/m2 of romidepsin
  Interventions: Drug: FK228 (romidepsin)

INTERVENTIONS:
Drug: FK228 (romidepsin) — Patients receive 13 mg/m2 of romidepsin (FK228) intravenously over 4 hours on Days 1, 8, and 15 of each 28-day cycle.
  Other Names: romidepsin

SUMMARY:
The purpose of this study is to evaluate the activity of FK228 in metastatic renal cell carcinoma (RCC) patients who have developed progressive disease (PD) following or during treatment with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all of the following criteria to be eligible for study participation:

* Age ≥ 18 years;
* Histologically confirmed Renal Cell Carcinoma (RCC);
* Metastatic disease, with measurable lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST);
* Failure of prior cytokine therapy;
* Documented progressive disease;

Exclusion Criteria:

Patients are ineligible for entry if any of the following criteria are met:

* Significant cardiac disease including congestive heart failure, history of myocardial infarction within one year, uncontrolled dysrhythmias, or poorly controlled angina
* History of serious ventricular arrhythmia
* Corrected QT interval (QTc) ≥ 500 msec
* Known infection with Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C;
* Previous extensive radiotherapy involving ≥ 30% of bone marrow
* Coexistent second malignancy or history of prior malignancy within previous 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-05-01 (Actual); Primary Completion 2004-08-01 (Actual); Study Completion 2004-08-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the rate of objective response (the best response of Complete Response (CR), Partial Response (PR)). | Up to 6 months

SECONDARY OUTCOMES:
Rate of disease control, Complete Response, Partial Response, or Stable Disease | Up to 6 months
Time to objective disease progression. | Up to 6 months
Number of Participants with Adverse Events | Up to 6 months
Change from screening assessment to the final study visit in Karnofsky performance status. | Up to 6 months
Steady state plasma concentrations | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: William McCulloch, MB, FRCP, Study Director — Gloucester Pharmaceuticals Inc.
Locations (3):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - University of Chicago, Chicago, Illinois
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Background] Moreno L, Casanova M, Chisholm JC, Berlanga P, Chastagner PB, Baruchel S, Amoroso L, Gallego Melcon S, Gerber NU, Bisogno G, Fagioli F, Geoerger B, Glade Bender JL, Aerts I, Bergeron C, Hingorani P, Elias I, Simcock M, Ferrara S, Le Bruchec Y, Slepetis R, Chen N, Vassal G. Phase I results of a phase I/II study of weekly nab-paclitaxel in paediatric patients with recurrent/refractory solid tumours: A collaboration with innovative therapies for children with cancer. Eur J Cancer. 2018 Sep;100:27-34. doi: 10.1016/j.ejca.2018.05.002. Epub 2018 Jun 21. PMID 29936064
- [Background] Wolchok J. Putting the Immunologic Brakes on Cancer. Cell. 2018 Nov 29;175(6):1452-1454. doi: 10.1016/j.cell.2018.11.006. PMID 30500529
- [Background] Mansfield AS, Jen J. Predicting Treatment Response Based on RNA Expression in Large Datasets. Clin Cancer Res. 2019 Mar 1;25(5):1443-1445. doi: 10.1158/1078-0432.CCR-18-2823. Epub 2018 Nov 16. PMID 30446588
- [Background] Pal SK, Forero-Torres A, Thompson JA, Morris JC, Chhabra S, Hoimes CJ, Vogelzang NJ, Boyd T, Bergerot PG, Adashek JJ, Li H, Yu X, Gartner EM, Carret AS, Smith DC. A phase 1 trial of SGN-CD70A in patients with CD70-positive, metastatic renal cell carcinoma. Cancer. 2019 Apr 1;125(7):1124-1132. doi: 10.1002/cncr.31912. Epub 2019 Jan 9. PMID 30624766
- [Background] Stadler W, et al. A phase II study of depsipeptide (Dep) in patients (pts) with metastatic renal cell cancer (RCC). J Clin Oncol. 2005 Jun; 23(16_suppl):4669.
- [Result] Stadler WM, Margolin K, Ferber S, McCulloch W, Thompson JA. A phase II study of depsipeptide in refractory metastatic renal cell cancer. Clin Genitourin Cancer. 2006 Jun;5(1):57-60. doi: 10.3816/CGC.2006.n.018. PMID 16859580